CLINICAL TRIAL: NCT01460446
Title: A Prospective, Multi-centre Study With Diabetic Patients Randomized to 24 Weeks Treatment Supported by Either Accu-Chek® Aviva Expert Blood Glucose Meter With an Integrated Bolus Advisor or MDI Standard Therapy With Accu-Chek® Aviva Nano Meter (Without Bolus Advisor)
Brief Title: ACCU-CHEK® Aviva Expert Study: Does Use of a Bolus Advisor Improve Glycemic Control in Patients Not Achieving Optimal Control Using Multiple Daily Injections (MDI)?
Acronym: ABACUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RD001333
Record Dates: First submitted 2011-09-22; First posted 2011-10-26 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-01

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

ARMS (2):
- Aviva Expert blood glucose meter (Experimental): Participants used the Accu-Chek® Aviva Expert blood glucose meter with an integrated bolus advisor to determine the dose of insulin for each injection in their 24 week multiple daily injection therapy.
  Interventions: Device: Aviva Expert blood glucose meter
- Aviva Nano blood glucose meter (Active Comparator): Participants used the Accu-Chek® Aviva Nano blood glucose meter and manual bolus calculation to determine the dose of insulin for each injection in their 24 week multiple daily injection therapy.
  Interventions: Device: Aviva Nano blood glucose meter

INTERVENTIONS:
Device: Aviva Expert blood glucose meter
  Arms: Aviva Expert blood glucose meter
Device: Aviva Nano blood glucose meter
  Arms: Aviva Nano blood glucose meter

SUMMARY:
This clinical, prospective, randomized, multi-center study determined if the use of an insulin bolus advisor improves glycemic control as measured by a change in HbA1c in patients failing multiple daily injection/intensified conventional therapy (MDI/ICT).

DETAILED DESCRIPTION:
Eligible participants were randomized to 24 weeks multiple daily injection therapy using either the Accu-Chek® Aviva Expert blood glucose meter with an integrated bolus advisor or the Accu-Chek® Aviva Nano blood glucose meter and manual bolus calculation.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older.
* Diagnosed with Type 1 or Type 2 diabetes.
* Recent HbA1c > 7.5% (measured within the last 6 weeks at local laboratory).
* On multiple daily injection (MDI) therapy for at least 6 months consisting of 1-2 injections per day of long-acting basal insulin (Lantus® or Detemir®) and at least 2 injections per day of regular or rapid-acting analog insulin for meal coverage.
* Subject adjusts meal insulin doses based on carbohydrate content of meals.
* Subject with Type 2 diabetes may be on stable metformin therapy (therapy unchanged during 3 months prior to study).
* Subject has been in Investigator's practice for at least 3 months but may have been seen by another physician in the practice.
* Subject has completed carbohydrate (CHO) training within the last 2 years.

Exclusion Criteria:

* Subject is on a therapy regimen that conflicts with the study:

  * Neutral protamine Hagedorn (NPH) or pre-mixed insulin;
  * oral anti-diabetic agents, with the exception of metformin;
  * injectable anti-diabetic agents other than long-acting insulin and rapid-acting insulin analogs or regular insulin (eg, fixed dose therapy);
  * use of sliding scale insulin therapy that determines insulin dosages based exclusively on specific blood glucose (bG) results.
* Subject has participated in another interventional trial within 6 weeks prior to study.
* Subject has been diagnosed with any clinically significant infectious disease or major organ system disease, such as gastroparesis or renal disease (at Investigator's discretion).
* Subject has used systemic oral or inhaled steroids for more than 7 days within the last 3 months.
* Subject is on chemotherapy or radiation therapy (self-reported).
* Subject is pregnant or lactating or is currently planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2011-10; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iris Vesper, Study Director — Roche Diagnostics GmbH
Locations (30):
- Germany (14):
  - Aschaffenburg
  - Augsburg
  - Berlin
  - Duisburg
  - Essen
  - Furth im Wald
  - Köln-Weiden
  - Leipzig
  - München
  - Münster
  - Rostock
  - Simmern
  - Unterhaching
  - Wurzen
- United Kingdom (16):
  - Blackburn
  - Bournemouth
  - Bradford
  - Chester
  - Cosham
  - Coventry
  - Derby
  - Exeter
  - Leicester
  - Lindley, Huddersfield
  - Middlesbrough
  - Northampton
  - Nottingham
  - Rotherham
  - Scunthorpe
  - Sheffield

REFERENCES:
- [Derived] Cavan DA, Ziegler R, Cranston I, Barnard K, Ryder J, Vogel C, Parkin CG, Koehler W, Vesper I, Petersen B, Wagner RS. Automated bolus advisor control and usability study (ABACUS): does use of an insulin bolus advisor improve glycaemic control in patients failing multiple daily insulin injection (MDI) therapy? [NCT01460446]. BMC Fam Pract. 2012 Oct 13;13:102. doi: 10.1186/1471-2296-13-102. PMID 23062116

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Started | 105 | 113
Completed | 100 | 93
Not Completed | 5 | 20
Not completed — Non-compliance | 2 | 9
Not completed — Consent Withdrawn | 0 | 4
Not completed — Non-compliance & Consent Withdrawn | 1 | 3
Not completed — Surgery/Illness | 1 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Other Reasons Incl. Lost for Follow-Up | 0 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter | Total
Number analyzed (Participants) | 105 | 113 | 218
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (13.5) | 42.0 (14.5) | 42.4 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 53 | 97
  Male | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin A1c (HbA1c) From Baseline to Week 24
Description: HbA1C was measured in blood samples at a central laboratory.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 100 | 93
Percentage | -0.66 (0.72) | -0.47 (0.70)

2. Secondary Outcome: Percentage of Blood Glucose Measurements Within the Blood Glucose Target Range From Screening to Baseline and From Week 23 to Week 24
Description: Participants measured their blood glucose at least 3-4 times daily throughout the study. The mean blood glucose level was calculated for each 3-day period from Baseline to Week 24 and the percentage of 3-day blood glucose levels with the target range of 70-180 mg/dL (3.9-10 mmol/L) was calculated for the 2 reporting periods of Screening to Baseline and Week 23 to Week 24.
Time Frame: Screening to Week 24
Population: Intent-to-treat population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: Percentage of measurements
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 100 | 93
Percentage of measurements
  Screening to Baseline (n=92, 86) | 50.6 (14.3) | 50.7 (15.1)
  Week 23 to Week 24 (n=92, 86) | 49.3 (17.2) | 52.2 (15.5)

3. Secondary Outcome: Number of Symptomatic Hypoglycemic Episodes Per Subject Year From Screening to Baseline and From Week 23 to Week 24
Description: A symptomatic hypoglycemic episode was defined as an event with symptoms consistent with hypoglycemia which was confirmed by a blood glucose reading < 70 mg/dL (3.9 mmol/L). Symptoms might include but were not limited to sweating, dizziness, lightheadedness, tremors, nervousness, hunger, headaches, and weakness or tiredness.
Time Frame: Screening to Week 24
Population: Intent-to-treat population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: Episodes per year
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 100 | 93
Episodes per year
  Screening to Baseline (n=100, 93) | 18.9 (50.8) | 23.2 (73.8)
  Week 23 to Week 24 (n=93, 91) | 17.0 (43.6) | 15.8 (56.7)

4. Secondary Outcome: Change in the Mean Amplitude of Glucose Excursion (MAGE) From Baseline to Week 24
Description: Approximately half of the investigational sites monitored glucose levels in participants enrolled in this study using the DexCom Seven® Plus Continuous Glucose Monitoring device. The device provides glucose measurements every 5 minutes for up to 7 days. The system contains a sensor, transmitter, and receiver. The sensor is a flexible round wire that goes under the skin to read glucose levels. The transmitter snaps into the sensor and wirelessly sends glucose readings to the receiver. Data was obtained from approximately one-third of participants and was used to calculate MAGE. Data were collected in the 3 days prior to Baseline and the Week 24 visit. The standard deviation of the blood glucose measurements in each 3-day period was calculated. For each glucose measurement, the difference from the previous reading was calculated. Absolute differences smaller than the standard deviation were discarded. MAGE is the mean of the remaining difference scores.
Time Frame: 3 days prior to Baseline to Week 24
Population: Intent-to-treat population: All randomized participants with continuous glucose monitoring data at Baseline and at Week 24 who completed the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 34 | 35
mg/dL | -20.2 (41.1) | -2.9 (32.1)

5. Secondary Outcome: Percentage of Bolus Opportunities Where the Accu-Chek® Aviva Expert Blood Glucose Meter Bolus Advisor Was Used During the Study
Description: Participants using the Accu-Chek® Aviva Expert blood glucose meter were encouraged to use the Bolus Advisor utility incorporated into the meter. A bolus opportunity occurs, for example, just before eating a meal.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants.
Measure: Mean (Standard Deviation); unit: Percentage of opportunities
Arm/Group | Aviva Expert Blood Glucose Meter
Number analyzed (Participants) | 105
Percentage of opportunities | 73.5 (21.9)

6. Secondary Outcome: Number of Accu-Chek® Aviva Expert Blood Glucose Meter Bolus Advices Modified Per Day by Participants During the Study
Description: as for outcome 5
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants.
Measure: Mean (Standard Deviation); unit: Number of advices modified per day
Arm/Group | Aviva Expert Blood Glucose Meter
Number analyzed (Participants) | 105
Number of advices modified per day | 0.3 (0.5)

7. Secondary Outcome: Correct and Incorrect Use of Insulin:Carbohydrate Ratio (I:CHO) and Insulin Sensitivity Factor (ISF) Advice by Participants Using the Aviva Nano Blood Glucose Meter During the Study
Description: Participants using the Aviva Nano blood glucose meter received individualized advice in how to use their insulin:carbohydrate ratio (I:CHO) and insulin sensitivity factor (ISF) values to determine their insulin dose. The I:CHO ratio advice was considered to have been used correctly if the meal bolus dose the participant indicated in his/her patient diary was in accordance with the dose which could be calculated based upon the participant's total carbohydrate intake and the I:CHO ratio. The ISF advice was considered to have been correctly used if the correction bolus dose the participant indicated in his/her patient diary was in accordance with the dose which could be calculated based upon the participant's blood glucose target, current blood glucose value, and the ISF.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants who completed the study. Results are only reported for participants using the Aviva Nano blood glucose meter who had data available for analysis.
Measure: Mean (Standard Deviation); unit: Number of advices per day
Arm/Group | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 88
Number of advices per day
  I:CHO - correct (n=88) | 1.55 (1.1)
  I:CHO - incorrect (n=88) | 1.77 (0.9)
  ISF - correct (n=78) | 0.81 (0.7)
  ISF - incorrect (n=78) | 2.14 (0.9)

8. Secondary Outcome: Change in Carbohydrate Counting Accuracy From Baseline to Week 24
Description: Participants were asked to assess the carbohydrate content (grams) of 10 standardized meals by using a set of Dose Adjustment for Normal Eating (DAFNE) plates, which provide standardized photographs of meals with known carbohydrate values. The mean meal error (MME), an indicator of accuracy, and mean meal absolute error (MMAE), an indicator of variability were calculated from their responses. The MME is defined as the mean of the differences between the estimated carbohydrate content and the actual carbohydrate content over the 10 DAFNE plates. A negative MME indicates an underestimation and a positive MME indicates an overestimation of the actual carbohydrate content. The MMAE is defined as the mean of the absolute value of the differences between the estimated carbohydrate content and the actual carbohydrate content over the 10 DAFNE plates. The MMAE is ≥ 0 with a lower value indicating a better ability to estimate the actual carbohydrate content.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants who completed the study and had data available for analysis.
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 99 | 92
Grams
  Mean Meal Error | -0.90 (10.0) | 0.07 (11.2)
  Mean Meal Absolute Error | -2.9 (8.2) | 0.9 (9.4)

9. Secondary Outcome: Change in the Patient Health Questionnaire Depression Scale (PHQ-8) Score From Baseline to Week 24
Description: The Patient Health Questionnaire depression scale (PHQ-8) contains 8 items which can be rated from 0='not at all' to 3='nearly every day'. The total PHQ-8 score is the sum of the responses to the 8 items and ranges from 0 to 24. A lower score indicates less depression. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants who had data available for analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 95 | 89
Units on a scale | -0.36 (3.21) | -0.08 (3.87)

10. Secondary Outcome: Number of Participants With None, Mild, Moderate, Moderately Severe, and Severe Depression at Baseline and Week 24
Description: The Major Depression Disorder (MDD) scale is derived from the Patient Health Questionnaire depression scale (PHQ-8) and was used to categorize participants in regard to the severity of their depression. There are 5 categories on the MDD scale: None, mild, moderate, moderately severe, and severe. The category for each participant is determined from their PHQ-8 score. A total PHQ-8 score of 0 to 4 represents no significant depressive symptoms. A total PHQ-8 score of 5 to 9 represents mild depressive symptoms; 10 to 14, moderate; 15 to 19, moderately severe; and 20 to 24, severe. A higher score indicates more depression.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants who completed the study.
Measure: Number; unit: Participants
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 100 | 93
Participants
  Baseline - None (n=100, 93) | 66 | 55
  Baseline - Mild (n=100, 93) | 22 | 26
  Baseline - Moderate (n=100, 93) | 11 | 9
  Baseline - Moderately Severe (n=100, 93) | 1 | 2
  Baseline - Severe (n=100, 93) | 0 | 1
  Week 24 - None (n=95, 89) | 67 | 54
  Week 24 - Mild (n=95, 89) | 21 | 23
  Week 24 - Moderate (n=95, 89) | 7 | 10
  Week 24 - Moderately Severe (n=95, 89) | 0 | 2
  Week 24 - Severe (n=95, 89) | 0 | 0

11. Secondary Outcome: Change in the Problem Area in Diabetes (PAID) Scale Score From Baseline to Week 24
Description: The Problem Area in Diabetes (PAID) scale contains 20 items which can be rated from 0='not a problem' to 4='serious problem'. The total PAID scale score ranges from 0 to 80 with a higher score indicating more diabetes-related problems. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants who completed the study and had data available for analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 97 | 91
Units on a scale | -4.4 (11.2) | -4.4 (8.6)

12. Secondary Outcome: Change in the Hypoglycemia Fear Survey (HFS-II) Score From Baseline to Week 24
Description: The Hypoglycemia Fear Survey-II (HFS-II) contains 33 items (15 items regarding behavior and 18 items regarding worry) which can be rated from 0='never' to 4='always'). The total HFS-II score ranges from 0 to 132 with a higher score indicating more fear. A negative change score indicates improvement.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants who completed the study and had data available for analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 97 | 91
Units on a scale | -3.7 (13.3) | -5.9 (11.9)

13. Secondary Outcome: The Diabetes Treatment Satisfaction Questionnaire at Baseline (DTSQs) Score and the Diabetes Treatment Satisfaction Questionnaire for Change From Baseline (DTSQc) Score
Description: The Diabetes Treatment Satisfaction Questionnaire at Baseline (DTSQs) contains 6 items which can be scored from 0='very bad' to 6='very good'. The total score is the sum of the scores of the 6 items and ranges from 0 to 36. A higher score indicates more satisfaction. This questionnaire was administered at Baseline only.
  The Diabetes Treatment Satisfaction Questionnaire for change from Baseline (DTSQc) to study end contains 6 items which can be rated from -3='much worse now' to 3='much better now'). The total score is the sum of the scores of the 6 items and ranges from -18 to 18. A higher score indicates more satisfaction. This questionnaire was administered at the end of the study (Week 24) only.
Time Frame: Baseline to Week 24
Population: Intent-to-treat population: All randomized participants who completed the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Number analyzed (Participants) | 100 | 93
Units on a scale
  Baseline (n=99, 93) | 27.9 (6.2) | 28.1 (5.7)
  Week 24 (n=98, 92) | 11.4 (6.0) | 8.9 (6.3)

ADVERSE EVENTS:
Description: Intent-to-treat population: All randomized participants.
Arm/Group | Aviva Expert Blood Glucose Meter | Aviva Nano Blood Glucose Meter
Serious Adverse Events (participants affected / at risk) | 8/105 | 10/113
Other Adverse Events (participants affected / at risk) | 49/105 | 56/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aviva Expert Blood Glucose Meter (N=105) | Aviva Nano Blood Glucose Meter (N=113)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1
Urinary tract infection viral (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Tracheal injury (Injury, poisoning and procedural complications) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Change of bowel habit (Gastrointestinal disorders) | 1 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aviva Expert Blood Glucose Meter (N=105) | Aviva Nano Blood Glucose Meter (N=113)
Hypoglycaemia (Metabolism and nutrition disorders) | 44 | 34
Nasopharyngitis (Infections and infestations) | 15 | 30
Diarrhoea (Gastrointestinal disorders) | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.